CLINICAL TRIAL: NCT02525692
Title: Oral ONC201 in Adult Recurrent Glioblastoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The Sponsor terminated the study to prioritize enrollment in a randomized Phase 3 trial of ONC201 in an earlier setting. This decision was unrelated to any safety concerns with dordaviprone (ONC201).
Sponsor: Jazz Pharmaceuticals (Industry)
Collaborators: Oncoceutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ONC006
Record Dates: First submitted 2015-08-14; First posted 2015-08-17 (Estimated); Results first posted 2024-12-24 (Actual); Last update posted 2024-12-24 (Actual); Status verified 2024-12

CONDITIONS: Glioblastoma; Diffuse Midline Glioma; H3 K27M Glioma; Thalamic Glioma; Infratentorial Glioma; Basal Ganglia Glioma
MeSH Terms: conditions — Glioblastoma | interventions — TIC10 compound

ARMS (6):
- Arm A (Experimental): Patients had histologically confirmed World Health Organization Grade IV glioblastoma with any number of recurrences.
  Patients received 625 mg dordaviprone (ONC201) once every 3 weeks.
  Interventions: Drug: Dordaviprone (ONC201)
- Arm B (Experimental): Patients had first recurrence histologically confirmed World Health Organization Grade IV glioma.
  Patients received 625 mg dordaviprone (ONC201) weekly (Days 1, 8, and 15 of each cycle).
  Interventions: Drug: Dordaviprone (ONC201)
- Arm C (Experimental): Patients had clinical and/or radiographic evidence of first recurrence of histologically confirmed World Health Organization Grade IV glioblastoma and were eligible for salvage surgical resection.
  Patients received 625 mg dordaviprone (ONC201) weekly (Days 1, 8, and 15 of each cycle). Surgical resection was performed approximately 24 hours after at least the second dose of ONC201.
  Interventions: Drug: Dordaviprone (ONC201)
- Arm D (Experimental): Patients had confirmed World Health Organization Grade IV glioma with H3 K27M mutation (any number of recurrences were allowed).
  Patients received 625 mg dordaviprone (ONC201) weekly (Days 1, 8, and 15 of each cycle).
  Interventions: Drug: Dordaviprone (ONC201)
- Arm E (Experimental): Patients had clinical and/or radiographic evidence of midline glioma (recurrent disease was not required) and were eligible for salvage surgical resection.
  Patients received 625 mg dordaviprone (ONC201) weekly (Days 1, 8, and 15 of each cycle). Surgical resection was performed approximately 24 hours after at least the second dose of dordaviprone (ONC201).
  Interventions: Drug: Dordaviprone (ONC201)
- Arm F (Experimental): Patients had diffuse midline glioma involving the brainstem, thalamus, or spinal cord, without the H3 K27M mutation or with unknown H3 mutation status.
  Patients received 625 mg dordaviprone (ONC201) weekly (Days 1, 8, and 15 of each cycle).
  Interventions: Drug: Dordaviprone (ONC201)

INTERVENTIONS:
Drug: Dordaviprone (ONC201) — Dordaviprone (ONC201) is a brain-penetrant, small-molecule imipridone that acts as a mitochondrial caseinolytic protease P (ClpP) agonist and a dopamine receptor D2 (DRD2) antagonist.
  Other Names: Dordaviprone

SUMMARY:
This was a Phase 2, open-label, 6-arm, multi-center study of dordaviprone (ONC201) in patients with recurrent glioblastoma (Arms A, B, and C), H3 K27M-mutant diffuse glioma (Arm D), or diffuse midline glioma (Arms E and F).

The primary objective of this study was the assessment of dordaivprone (ONC201) anti-tumor activity through progression-free survival at 6 months using Response Assessment in Neuro-Oncology (RANO) criteria for high-grade glioma (HGG).

DETAILED DESCRIPTION:
This study included 6 arms:

* Patients in Arm A received 625 mg oral dordaviprone (ONC201) every 3 weeks.
* Patients in Arms B, C, D, E, and F received 625 mg oral dordaviprone (ONC201) every 1 week (Days 1, 8 and 15 of each cycle).
* Patients in Arms C and E received salvage surgical resection of their brain tumor 1 day after the second (or more) dose of dordaviprone (ONC201).

All patients underwent clinical evaluation after each cycle (defined as every 3 weeks).

Neuroimaging studies (contrast-enhanced brain magnetic resonance imaging or computed tomography for patients unable to undergo MRI) were performed at baseline, 8 weeks from treatment initiation, and then every 8 weeks thereafter.

Assessments of dordaviprone (ONC201) anti-tumor activity were assessed through progression-free survival at 6 months using RANO-HGG criteria. Safety was assessed through the reporting of adverse events, measurement of vital signs, electrocardiograms, and clinical laboratory results.

This study was terminated by an administrative protocol amendment (17 January 2023). The decision to terminate the study was not related to any safety concerns with dordaviprone (ONC201). Before the study was terminated, a total of 84 patients were enrolled and received at least 1 dose of dordaviprone (ONC201).

ELIGIBILITY:
Inclusion Criteria:

A patient had to meet all of the following criteria to be eligible to participate in the study:

1. For Arms A, B, and C: Had histologically confirmed World Health Organization (WHO) Grade IV glioblastoma. For Arm D: Must have had a WHO Grade IV glioma and the tumor must have harbored a histone H3 K27M mutation detected in a Clinical Laboratory Improvement Amendment (CLIA) certified laboratory by immunohistochemistry or DNA sequencing test on any glioma tumor sample. The H3 K27M mutation was often reported as H3 K28M in gene sequencing assays. For Arm E: Must have had clinical and/or radiographic evidence of a midline glioma (involving the brainstem, thalamus, spinal cord, hypothalamus, basal ganglia, brainstem [non-diffuse intrinsic pontine glioma (DIPG)], cerebellum, cerebellar peduncle, midline cortex, corpus collosum, pineal region, optic tract, or optic chiasm), and was eligible for salvage surgical resection as deemed by the site Investigator. For Arm F: Must have had a diffuse midline glioma that involved the brainstem, thalamus, or spinal cord, without the H3 K27M mutation or with unknown H3 mutation status at the time of enrollment.
2. Had unequivocal evidence of progressive disease on contrast-enhanced brain computed tomography (CT) or magnetic resonance imaging (MRI) as defined by Response Assessment in Neuro-Oncology (RANO) high-grade glioma (HGG) criteria, or had documented recurrent glioblastoma or WHO Grade IV glioma on diagnostic biopsy. For Arm E, patients were not required to have evidence of recurrent disease for inclusion.
3. Had previous first line therapy with at least radiotherapy and temozolomide. For patients who had tumors that exhibited unmethylated MGMT promoter, prior treatment with temozolomide was not required. For Arms D, E, and F: Must have had previous first line therapy with at least radiotherapy.
4. For Arm A and D: Any number of recurrences were allowable. For Arm B: Must have been first recurrence (only) WHO Grade IV glioma. First recurrence was defined as the progression following initial therapy (i.e., radiation ±chemotherapy). For patients who had prior therapy with radiation or chemotherapy for a low-grade glioma (LGG), the surgical diagnosis of the HGG was considered the first recurrence. For patients who did not receive additional treatment following surgery and diagnosis of the LGG, surgical diagnosis of HGG was not considered the first recurrence. Instead, progression after treatment was considered first recurrence. For Arm C: Patients must have had clinical and/or radiographic evidence of first recurrence of glioblastoma and must have been eligible for salvage surgical resection as deemed by the site Investigator. For Arm E: Recurrent disease was not required. Patients must have had a midline glioma, and must have been eligible for salvage surgical resection as deemed by the site Investigator.
5. Had an interval of at least 90 days from the completion of radiotherapy to the first dose of ONC201. If patients were within 90 days of radiotherapy, then the progressive lesion must have been outside of the high-dose radiation target volume or must have had unequivocal evidence of progressive tumor on a biopsy specimen.
6. From the projected start of scheduled study treatment, the following time periods must have elapsed: 5 half-lives from any investigational agent, 4 weeks from cytotoxic therapy (except 23 days for temozolomide and 6 weeks from nitrosoureas), 6 weeks from antibodies, or 4 weeks (or 5 half-lives, whichever was shorter) from other anti-tumor therapies.
7. All adverse events Grade >1 related to prior therapies (chemotherapy, radiotherapy, and/or surgery) must have been resolved, except for alopecia.
8. Were male or female aged ≥16 years.
9. Had a Karnofsky Performance Status (KPS) of ≥60.
10. Had adequate organ and marrow function as defined below; all screening labs should have been performed within 14 days of treatment initiation:

    * leukocytes: ≥3,000/mcL
    * absolute neutrophil count: ≥1,500/mcL
    * platelets: ≥100,000/mcL
    * hemoglobin: >8.0 mg/dL
    * total bilirubin: <2.0 × upper limit of normal (ULN)
    * aspartate aminotransferase/alanine aminotransferase (SGOT)/(SGPT): ≤2.5 × ULN
    * creatinine: ≤ULN OR
    * creatinine clearance: ≥60 mL/min/1.73 m2 for patients who had creatinine levels above normal.
11. Had a CT or MRI within 14 days prior to start of study drug.
12. Corticosteroid dose must have been stable or decreasing for at least 5 days prior to the baseline CT or MRI scan. For Arm B: Corticosteroid dose must have been stable or decreasing for at least 2 weeks prior to study entry.
13. The effects of ONC201 on the developing human fetus are unknown. For this reason, women of childbearing potential and men must have agreed to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Should a woman have become pregnant or suspected that she was pregnant while she or her partner were participating in this study, she should have informed her treating physician immediately. Male subjects should have agreed to use adequate method of contraception starting with the first dose of study therapy through 120 days after the last dose of therapy.
14. Had archival tissue for evaluation of correlative objectives (if available). Archival tissue was required for Arms B and C.
15. Had the ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

A potential patient who met any of the following criteria was ineligible to participate in the study:

1. Had a history of allergic reactions attributed to compounds of similar chemical or biologic composition to ONC201 or its excipients.
2. Had current or planned participation in a study of an investigational agent or using an investigational device.
3. Had uncontrolled intercurrent illness including, but not limited to, ongoing or active infection or psychiatric illness/social situations that would have limited compliance with study requirements.
4. Had an active infection that required systemic therapy.
5. Patients who had prior stereotactic radiotherapy, convection enhanced delivery (CED) or brachytherapy must have had a biopsy to confirm radiographic progression was consistent with progressive tumor and not treatment-related necrosis. If the recurrent lesion was outside of any prior high-dose radiation target volume or distant from the prior CED or brachytherapy site, patients were considered eligible
6. Was a pregnant woman because ONC201 is novel agent with unknown potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with ONC201, breastfeeding should have been discontinued if the mother was treated with ONC201.
7. Had known human immunodeficiency virus (HIV)-positive test on combination antiretroviral therapy.
8. Had a known history of cardiac arrhythmias including atrial fibrillation, tachyarrhythmias or bradycardia. Patients who were receiving therapeutic agents known to prolong QT interval were excluded. Patients who had a history of congestive heart failure, myocardial infarction, or stroke within the last 3 months were excluded.
9. Had active illicit drug use or diagnosis of alcoholism.
10. For Arms A, B, and C: Had prior bevacizumab treatment (this prior treatment was allowable for patients in Arms D, E, and F).
11. Had tumors with known isocitrate dehydrogenase 1 (IDH1) or known IDH2 mutations as determined by immunohistochemistry for the IDH1 R132H variant or by direct sequencing.
12. Had any known additional malignancies that were progressing or required active treatment within 3 years of start of study drug. Exceptions included basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or in situ cervical cancer that had undergone potentially curative therapy.
13. Had undergone any surgery (not including minor diagnostic procedures such as lymph node biopsy) within 2 weeks of baseline disease assessments; or were not fully recovered from any side effects of previous procedures.
14. Had concomitant use of cytochrome P450 (CYP)3A4/5 inhibitors during the treatment phase of the study and within 72 hours prior to starting study drug administration.
15. Had concomitant use of potent CYP3A4/5 inducers, which included enzyme inducing antiepileptic drugs (EIAEDs), during the treatment phase of the study and within 2 weeks prior to starting treatment.
16. Had planned concurrent use Optune™. Prior use of the device was allowable.
17. For Arms D and F: Had evidence of leptomeningeal spread of disease.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2023-04-17 (Actual); Study Completion 2023-04-17 (Actual)

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - University of California, Los Angeles, Los Angeles, California
  - Miami Cancer Institute, Miami, Florida
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - University of Utah, Huntsman Cancer Institute, Salt Lake City, Utah

REFERENCES:
- [Derived] Arrillaga-Romany I, Gardner SL, Odia Y, Aguilera D, Allen JE, Batchelor T, Butowski N, Chen C, Cloughesy T, Cluster A, de Groot J, Dixit KS, Graber JJ, Haggiagi AM, Harrison RA, Kheradpour A, Kilburn LB, Kurz SC, Lu G, MacDonald TJ, Mehta M, Melemed AS, Nghiemphu PL, Ramage SC, Shonka N, Sumrall A, Tarapore RS, Taylor L, Umemura Y, Wen PY. ONC201 (Dordaviprone) in Recurrent H3 K27M-Mutant Diffuse Midline Glioma. J Clin Oncol. 2024 May 1;42(13):1542-1552. doi: 10.1200/JCO.23.01134. Epub 2024 Feb 9. PMID 38335473
- [Derived] Weissenrieder JS, Reed JL, Moldovan GL, Johnson MT, Trebak M, Neighbors JD, Mailman RB, Hohl RJ. Antipsychotic drugs elicit cytotoxicity in glioblastoma multiforme in a calcium-dependent, non-D2 receptor-dependent, manner. Pharmacol Res Perspect. 2021 May;9(3):e00689. doi: 10.1002/prp2.689. PMID 34003586
- [Derived] Chi AS, Tarapore RS, Hall MD, Shonka N, Gardner S, Umemura Y, Sumrall A, Khatib Z, Mueller S, Kline C, Zaky W, Khatua S, Weathers SP, Odia Y, Niazi TN, Daghistani D, Cherrick I, Korones D, Karajannis MA, Kong XT, Minturn J, Waanders A, Arillaga-Romany I, Batchelor T, Wen PY, Merdinger K, Schalop L, Stogniew M, Allen JE, Oster W, Mehta MP. Pediatric and adult H3 K27M-mutant diffuse midline glioma treated with the selective DRD2 antagonist ONC201. J Neurooncol. 2019 Oct;145(1):97-105. doi: 10.1007/s11060-019-03271-3. Epub 2019 Aug 27. PMID 31456142

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm A: Patients with histologically confirmed WHO Grade IV glioblastoma with any number of recurrences.
  Patients received 625 mg oral ONC201 once every 3 weeks.
- Arm B: Patients with first recurrence of histologically confirmed WHO Grade IV glioma.
  Patients received 625 mg oral ONC201 once every week (Days 1, 8, and 15 of each cycle).
- Arm C: Patients with clinical and/or radiographic evidence of first recurrence of histologically confirmed WHO Grade IV glioblastoma and were eligible for salvage surgical resection.
  Patients received 625 mg oral ONC201 once weekly (Days 1, 8 and 15 of each cycle). Surgical resection was performed approximately 24 hours after at least the second dose of ONC201.
- Arm D: Patients with confirmed WHO Grade IV glioma with H3 K27M mutation (any number of recurrences were allowed).
  Patients received 625 mg oral ONC201 once weekly (Days 1, 8, and 15 of each cycle).
- Arm E: Patients with clinical and/or radiographic evidence of midline glioma (recurrent disease was not required) and were eligible for salvage surgical resection.
  Patients received 625 mg oral ONC201 once weekly (Days 1, 8 and 15 of each cycle). Surgical resection was performed approximately 24 hours after at least the second dose of ONC201.
- Arm F: Patients with diffuse midline glioma involving the brainstem, thalamus, or spinal cord, without H3 K27M mutation or with unknown H3 mutation status.
  Patients received 625 mg oral ONC201 once weekly (Days 1, 8, and 15 of each cycle).
Period: Overall Study
Arm/Group | Arm A | Arm B | Arm C | Arm D | Arm E | Arm F
Started | 17 | 19 | 8 | 30 | 3 | 7
Completed | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 17 | 19 | 8 | 30 | 3 | 7
Not completed — Withdrawal by Subject | 1 | 1 | 0 | 5 | 0 | 1
Not completed — Death | 16 | 18 | 7 | 20 | 3 | 6
Not completed — Lost to Follow-up | 0 | 0 | 1 | 5 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A | Arm B | Arm C | Arm D | Arm E | Arm F | Total
Number analyzed (Participants) | 17 | 19 | 8 | 30 | 3 | 7 | 84
Age, Continuous [Median (Full Range); unit: years] | 58.0 [22 to 74] | 56.0 [21 to 75] | 66.5 [48 to 80] | 35.0 [17 to 53] | 37.0 [26 to 40] | 50.0 [30 to 60] | 48.0 [17 to 80]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 10 | 6 | 14 | 1 | 4 | 43
  Male | 9 | 9 | 2 | 16 | 2 | 3 | 41
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1 | 5 | 0 | 0 | 7
  Not Hispanic or Latino | 16 | 17 | 7 | 22 | 3 | 7 | 72
  Unknown or Not Reported | 1 | 1 | 0 | 3 | 0 | 0 | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 2 | 0 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 1 | 0 | 1 | 0 | 2
  White | 15 | 18 | 7 | 24 | 2 | 6 | 72
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 2 | 1 | 0 | 4 | 0 | 0 | 7
Primary Tumor Location [Count of Participants; unit: Participants]
  Brainstem | 1 | 3 | 0 | 6 | 1 | 1 | 12
  Midline ex-brainstem | 3 | 3 | 1 | 17 | 2 | 6 | 32
  Non-midline | 13 | 13 | 7 | 7 | 0 | 0 | 40

OUTCOME MEASURES:

1. Primary Outcome: Percent of Patients With Probability of Progression-Free Survival at 6 Months
Description: Progression-free survival rate at 6 months was defined as the percentage of patients who exhibit progression-free survival for >6 months.
Time Frame: Progression-free survival assessments were conducted 6 months following treatment initiation.
Population: Note: In Arm B, one participant with recurrent H3 K27M-mutant glioblastoma and non-measurable disease experienced complete regression of enhancing lesions for >1.5 years was censored from analysis due to use of anastrozole at baseline and throughout the study.
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Arm A | Arm B | Arm C | Arm D | Arm E | Arm F
Number analyzed (Participants) | 17 | 19 | 8 | 30 | 3 | 7
percentage of patients | 11.8 [2.0 to 31.2] | 0 [NA to NA] — Not calculated due to insufficient number of participants with events. | NA [NA to NA] — Not calculated. By design, all patients in this cohort had surgery shortly after initiation of dordaviprone (ONC201) with no preceding post-baseline assessment; hence, all patients are censored for PFS at baseline. | 14.5 [4.6 to 29.8] | 0 [NA to NA] — Not calculated due to insufficient number of participants with events. | 14.3 [0.7 to 46.5]

ADVERSE EVENTS:
Time Frame: From the time/date of initiation of study treatment through 30 days following cessation of study treatment and prior to initiation of other anticancer therapy, up to a maximum of 87.2 months.
Arm/Group | Arm A | Arm B | Arm C | Arm D | Arm E | Arm F
All-Cause Mortality (participants affected / at risk) | 16/17 | 18/19 | 7/8 | 20/30 | 3/3 | 6/7
Serious Adverse Events (participants affected / at risk) | 6/17 | 1/19 | 1/8 | 11/30 | 1/3 | 1/7
Other Adverse Events (participants affected / at risk) | 16/17 | 17/19 | 5/8 | 29/30 | 2/3 | 7/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A (N=17) | Arm B (N=19) | Arm C (N=8) | Arm D (N=30) | Arm E (N=3) | Arm F (N=7)
Bradycardia (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0
Anal incontinence (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Disease progression (General disorders) | 2 | 0 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 1 | 0 | 0 | 1 | 0 | 0
Gait disturbance (General disorders) | 1 | 0 | 0 | 0 | 0 | 0
Chest pain (General disorders) | 0 | 0 | 0 | 1 | 0 | 0
Hypersensitivity (Immune system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 2 | 1 | 0
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0
Clavicle fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1
Troponin T increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0
Failure to thrive (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0
Tumor haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0
Headache (Nervous system disorders) | 0 | 0 | 1 | 2 | 0 | 0
Seizure (Nervous system disorders) | 3 | 0 | 0 | 1 | 0 | 0
Hemiparesis (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Brain oedema (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Cerebral haemorrhage (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Dysarthria (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Encephalopathy (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Hydrocephalus (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Intraventricular haemorrhage (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Urinary incontinence (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Hypopnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Pulmonary infarction (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A (N=17) | Arm B (N=19) | Arm C (N=8) | Arm D (N=30) | Arm E (N=3) | Arm F (N=7)
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 6 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 1 | 0 | 1 | 0 | 0
Leukopenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Bradycardia (Cardiac disorders) | 1 | 0 | 0 | 1 | 0 | 0
Atrioventricular block (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0
Sinus bradycardia (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0
Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1
Ear discomfort (Ear and labyrinth disorders) | 0 | 1 | 0 | 0 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 1
Cushingoid (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 1
Diplopia (Eye disorders) | 0 | 0 | 0 | 2 | 0 | 0
Vision blurred (Eye disorders) | 0 | 0 | 0 | 2 | 0 | 0
Dry eye (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1
Photophobia (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 5 | 3 | 1 | 7 | 0 | 4
Vomiting (Gastrointestinal disorders) | 1 | 2 | 1 | 5 | 0 | 2
Diarrhoea (Gastrointestinal disorders) | 1 | 3 | 0 | 4 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 2 | 0 | 3 | 1 | 1
Anal incontinence (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 0 | 1
Constipation (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0 | 0
Dry mouth (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 0 | 0
Toothache (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 6 | 4 | 0 | 5 | 0 | 2
Gait disturbance (General disorders) | 2 | 3 | 0 | 0 | 0 | 1
Oedema peripheral (General disorders) | 1 | 1 | 0 | 1 | 0 | 0
Asthenia (General disorders) | 0 | 0 | 0 | 1 | 1 | 0
Disease progression (General disorders) | 2 | 0 | 0 | 0 | 0 | 0
Hypersensitivity (Immune system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 1
Bronchitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Tinea pedis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 4 | 0 | 3 | 1 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1
Lymphocyte count decreased (Investigations) | 0 | 1 | 0 | 4 | 0 | 0
Neutrophil count decreased (Investigations) | 0 | 1 | 0 | 1 | 0 | 2
Platelet count decreased (Investigations) | 0 | 2 | 0 | 2 | 0 | 0
Alanine aminotransferase increased (Investigations) | 1 | 0 | 0 | 2 | 0 | 0
Blood alkaline phosphatase increased (Investigations) | 1 | 2 | 0 | 0 | 0 | 0
White blood cell count increased (Investigations) | 1 | 0 | 0 | 2 | 0 | 0
Blood glucose increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 1
Blood lactate dehydrogenase increased (Investigations) | 1 | 0 | 0 | 1 | 0 | 0
Blood phosphorus decreased (Investigations) | 1 | 1 | 0 | 0 | 0 | 0
Electrocardiogram QT prolonged (Investigations) | 0 | 0 | 0 | 1 | 0 | 1
Neutrophil count increased (Investigations) | 1 | 0 | 0 | 1 | 0 | 0
SARS-CoV-2 test positive (Investigations) | 0 | 0 | 0 | 2 | 0 | 0
Weight decreased (Investigations) | 1 | 0 | 0 | 1 | 0 | 0
Weight increased (Investigations) | 1 | 0 | 0 | 1 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0
Blood magnesium decreased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 3 | 4 | 1 | 4 | 0 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 5 | 1 | 0 | 3 | 1 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 5 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 2 | 1 | 0 | 3 | 0 | 0
Hypernatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 3 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1 | 0 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1 | 0 | 0
Failure to thrive (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0
Hyperphosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 4 | 1 | 2 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 2 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 3 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 2 | 0 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0
Headache (Nervous system disorders) | 2 | 5 | 2 | 8 | 1 | 1
Hemiparesis (Nervous system disorders) | 4 | 2 | 0 | 7 | 0 | 2
Seizure (Nervous system disorders) | 5 | 2 | 0 | 1 | 0 | 0
Aphasia (Nervous system disorders) | 3 | 3 | 0 | 1 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 3 | 0 | 4 | 0 | 0
Paraesthesia (Nervous system disorders) | 2 | 1 | 0 | 2 | 0 | 1
Dysarthria (Nervous system disorders) | 1 | 2 | 0 | 1 | 0 | 0
Hemianopia (Nervous system disorders) | 0 | 0 | 0 | 2 | 0 | 2
Memory impairment (Nervous system disorders) | 1 | 0 | 1 | 1 | 0 | 1
Somnlolence (Nervous system disorders) | 0 | 1 | 0 | 2 | 0 | 0
Brain oedema (Nervous system disorders) | 0 | 1 | 0 | 1 | 0 | 0
Haemorrhage intracranial (Nervous system disorders) | 2 | 0 | 0 | 0 | 0 | 0
Hypoaesthesia (Nervous system disorders) | 0 | 2 | 0 | 0 | 0 | 0
Tremor (Nervous system disorders) | 0 | 0 | 0 | 2 | 0 | 0
Apraxia (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Ataxia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Aura (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Balance disorder (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Cerebral haemorrhage (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Cognitive disorder (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Disturbance in attention (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Dysmetria (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Facial paresis (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Hemianaesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Syncope (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Vasogenic cerebral oedema (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Confusional state (Psychiatric disorders) | 2 | 2 | 0 | 2 | 0 | 0
Insomnia (Psychiatric disorders) | 1 | 2 | 0 | 0 | 0 | 0
Irritability (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 1
Depression (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0
Disorientation (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0
Urinary incontinence (Renal and urinary disorders) | 0 | 0 | 0 | 3 | 0 | 1
Dysuria (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1 | 0 | 1
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2 | 0 | 0
Dry throat (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Ingrowing nail (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Skin atrophy (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Skin discolouration (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 2 | 0 | 0 | 1 | 0 | 1
White blood cell count decreased (Investigations) | 0 | 0 | 0 | 1 | 0 | 2

LIMITATIONS AND CAVEATS:
The Sponsor terminated this study based on the initiation of a randomized, Phase 3 study of dordaviprone (ONC201) in an earlier setting; closing this study ensured that enrollment would not be competing against the Phase 3 study. The decision to terminate the study was not related to any safety concerns with dordaviprone (ONC201).

Note that at the time enrollment was halted, some treatment arms had not completed enrollment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Within 12 months of the completion of the Study at all sites, if no publication of the overall multi-center results has been made, institutions are entitled to publish their locally obtained results, provided the Sponsor is given the opportunity to review and comment. Institution publications may be delayed up to an additional 90 days to allow the Sponsor to seek patent protection.

DOCUMENTS (2):
  • Study Protocol (2021-06-03): https://cdn.clinicaltrials.gov/large-docs/92/NCT02525692/Prot_000.pdf
  • Statistical Analysis Plan (2023-05-24): https://cdn.clinicaltrials.gov/large-docs/92/NCT02525692/SAP_001.pdf